CLINICAL TRIAL: NCT07387705
Title: On Track for Wellness: Stepped-wedge Cluster Randomized Trial of a Fitbit Enhanced Health Intervention for Early Onset Psychosis
Brief Title: On Track for Wellness (OTW) Stepped Wedge Cluster Randomized Trial
Acronym: OTW
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STUDY2025-1399; HHS-2025-ACL-NIDILRR-RTHF-0123 (Other Grant/Funding Number: National Institute on Disability, Independent Living, and Rehabilitation Research (NIDILRR))
Record Dates: First submitted 2026-01-22; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Sleep; Physical Activity; First Episode Psychosis
Keywords: sleep; physical activity; first episode psychosis treatment
MeSH Terms: conditions — Motor Activity | interventions — Health

STUDY DESIGN:
Intervention Model Description: Stepped-wedge cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Services as Usual (No Intervention): Services as usual
- OTW intervention (Experimental): OTW intervention
  Interventions: Other: On Track for Wellness

INTERVENTIONS:
Other: On Track for Wellness — Client education regarding sleep and physical activity accompanied by use of a Fitbit tracker
  Arms: OTW intervention

SUMMARY:
This study will evaluate a program called On Track for Wellness (OTW) which is being adopted by the Illinois Department of Human Services' Division of Behavioral Health & Recovery (DBHR) for use in all state-funded early psychosis programs in Illinois. OTW combines use of Fitbit activity trackers with health education, goal setting to promote health activation, and ongoing support for maintaining healthy lifestyles. Successful completion of this research will gauge the effectiveness of this program in improving sleep hygiene and increasing physical activity among people recently diagnosed with schizophrenia or other psychotic disorders.

DETAILED DESCRIPTION:
The study involves 2 phases. The first phase involves a pilot test conducted in two of the state's 18 early psychosis programs, in which interview data will be gathered from 2 staff and 5 clients at each program (total N=4 staff and 10 clients). The second phase involves training all remaining programs to deliver OTW and using state administrative data as well as data from clients' Fitbit accounts to evaluate changes in client outcomes over the three-year study period.

ELIGIBILITY:
Inclusion Criteria: client at First Episode psychosis program -

Exclusion Criteria: not a client at a First Episode psychosis program

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 365 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2029-09-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Increase physical exercise | Day 1
  increase in # of steps per day

CONTACTS AND LOCATIONS:
Overall Officials: Judith A Cook, Ph.D, Principal Investigator — University of Illinois at Chicago

IPD SHARING:
Plan to Share IPD: No